CLINICAL TRIAL: NCT05161663
Title: Peer-driven Intervention Promoting PrEP Uptake Among African American and Hispanic/Latino MSM
Brief Title: Peer-driven Intervention on PrEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Rhode Island Public Health Institute (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1594759
Record Dates: First submitted 2021-08-26; First posted 2021-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: HIV Infections
Keywords: pre-exposure prophylaxis
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: This peer-driven intervention (PDI), modified based on respondent-driven sampling (RDS) or snowball sampling, is a "chain referral" approach. Index peers will be purposefully selected to reflect the diversity of African American (AA) and Hispanic/Latino (H/L) men who have sex with men (MSM) and are required to take a formal training about pre-exposure prophylaxis (PrEP) and HIV. These index peers will educate members of their social networks and encourage them to initiate PrEP. Those referred peers will schedule an appointment to complete a short survey and will be referred to our PrEP clinic if they are interested in PrEP uptake. The referred peers will serve as index peers for the following wave of recruitment. It is expected to achieve a robust sample of AA and H/L within six waves of recruitment. This PDI approach is potential to engage AA and H/L who are most at risk of HIV acquisition in PrEP uptake and could contribute to reducing the concentrated HIV epidemic.
Masking Description: No mask
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PDI group (Experimental): In this group, participants will receive education about HIV and pre-exposure prophylaxis (PrEP) and be referred to our study by peer educators. Referred participants will have free PrEP counseling and receive referrals if interested. We will follow up at three and six months and check participants' PrEP status.
  Interventions: Behavioral: Peer-driven intervention
- Control group (No Intervention): In the control group, participants do not receive any education from peers and will be directly recruited by research assistants from venues (e.g. gay bars, LGBTQ communities, LGBTQ events, and social media advertisements). Participants will receive PrEP counseling and referral if interested. We will follow up at three and six months and check participants' PrEP status.

INTERVENTIONS:
Behavioral: Peer-driven intervention — This peer-driven intervention (PDI), modified based on respondent-driven sampling (RDS) or snowball sampling, is a "chain referral" approach. Index peers will be purposefully selected to reflect the diversity of African American (AA) and Hispanic/Latino (H/L) men who have sex with men (MSM) and are required to take a formal training about pre-exposure prophylaxis (PrEP) and HIV. These index peers will educate members of their social networks and encourage them to initiate PrEP. Those referred peers will schedule an appointment to complete a short survey and will be referred to our PrEP clinic if they are interested in PrEP uptake. The referred peers will serve as index peers for the following wave of recruitment. It is expected to achieve a robust sample of AA and H/L within six waves of recruitment. This PDI approach is potential to engage AA and H/L who are most at risk of HIV acquisition in PrEP uptake and could contribute to reducing the concentrated HIV epidemic.
  Arms: PDI group

SUMMARY:
The objective of this study is to develop an effective peer-driven intervention (PDI) approach and assess its feasibility and efficacy on pre-exposure prophylaxis (PrEP) uptake among men who have sex with men.

DETAILED DESCRIPTION:
This proposed study aims to assess the effect of a peer-driven intervention (PDI) on promoting pre-exposure prophylaxis (PrEP) uptake among African American (AA) and Hispanic/Latino men who have sex with men (MSM). PDI is based on respondent-driven sampling (RDS) or snowball sampling. PDI is a chain referral approach and includes both peer referral and peer education. Index peers will be purposefully sampled to reflect the diversity of our study population through local clinics, community organizations, and online. Index peers will receive a four-hour formal training about PrEP and HIV, educate members of their social network, and encourage them to initiate PrEP. Each index peers will be given three referral coupons. Referred peers will schedule a research visit to complete a short survey and then be referred to the local PrEP clinic if they are interested in starting PrEP. These referred individuals will also serve as index peers for the following wave of recruitment. We expect to achieve a robust sample of AA and H/L MSM within six waves of recruitment as peers will educate and recruit study participants through their social networks.

Given the nature of RDS, the study design will include a concurrent non-randomized control group, which will be recruited using venue-based sampling (e.g. gay dance clubs, bars, and social organizations). This has been used in previous RDS studies as an appropriate study design and comparison group. We will identify appropriate venues that AA and H/L MSM frequent using one-to-one qualitative interviews in Specific Aim 1. Research staff will visit these venues at specific times to recruit AA and H/L MSM. MSM who are willing to participate in this study will receive PrEP and HIV education offered by research staff and complete a short survey during outreach. Individuals who are interested in PrEP uptake will be referred to the PrEP clinic. All study participants, regardless of PrEP status (initiated or not initiated), will be followed for six months. Each individual will complete three visits, including baseline, three-month, and six-month follow-ups.

This study has two independent arms. Our primary outcome is PrEP uptake, which is defined as a binary variable (Yes vs. No). We will calculate the study power using the method for two independent proportions power analyses. Our local STD clinic data shows only 8% of AA and H/L MSM have used PrEP and we will assume that 8% of AA and H/L MSM recruited through venue-based sampling will initiate PrEP. We expect to observe at least a 14% increase in PrEP uptake in the PDI group. To have 80% of power (Type I error =0.05), we will recruit 100 participants (N=100, 50 AA, and 50 H/L MSM) in each group.

PrEP uptake measured by receiving a prescription for the medication and filling a prescription at a pharmacy will be treated as time-to-event variables. We will perform survival analysis techniques (Kaplan-Meier models and Cox proportional hazards models) to assess the effect of the PDI on PrEP initiation. Self-reported PrEP adherence and drug concentration level (Yes vs. No) will be treated as binary variables and multivariate logistic regression will be performed.

ELIGIBILITY:
Eligibility Criteria 18 years of age or older Assigned male at birth and currently identify as male Having sex with men in the past three months Not currently on PrEP English- or Spanish-speaking

Exclusion Criteria:

Age less than 18 years, No having sex with men in the past 3 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2024-12-23 (Actual)

PRIMARY OUTCOMES:
Pre-exposure prophylaxis (PrEP) uptake | 0-6 months
  Self-report PrEP uptake
Pre-exposure prophylaxis (PrEP) persistence | 0-6 months
  the length of time on PrEP
Pre-exposure prophylaxis (PrEP) adherence | 0-6 months
  Self-reported medication adherence

CONTACTS AND LOCATIONS:
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data due to confidentiality considerations and the sensitive nature of behavioral and HIV-related information collected.